CLINICAL TRIAL: NCT04018261
Title: A Prospective Multicenter Open-label, Not Controlled Phase Ib-II Clinical Trial to Assess the Safety and Immunologic Efficacy of Virus-specific T Lymphocytes From the Best Donor in Receptors of Hematopoietic Progenitor Allogeneic Transplant
Brief Title: Virus-specific Activated T Lymphocytes From a Donor in Hematopoietic Progenitor Transplanted Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Vall d'Hebron Institute of Oncology (Other); Hospital Universitario La Fe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BST-LT-01
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: CMV Viremia; Immunosuppression-related Infectious Disease
Keywords: CMV; Bone marrow transplant; Activated T-Lymphocytes; Cell therapy; Virus infection; immunosuppression
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Activated T-Lymphocytes (Experimental): Allogeneic T-Lymphocytes obtained from apheresis activated against CMV.
  Interventions: Drug: Activated T-Lymphocytes

INTERVENTIONS:
Drug: Activated T-Lymphocytes — Activated T-Lymphocytes will be infused intravenously in a single-dose

SUMMARY:
Marrow transplanted immunocompromised patients with cytomegalovirus (CMV) viral infection will be treated with CMV activated T-Lymphocytes. T-Lymphocytes will be obtained through an apheresis from a compatible donor.

Safety and immunoreconstitution parameters in blood samples will be assessed up to +60 days after the treatment.

DETAILED DESCRIPTION:
A prospective, multicentre, open-label and uncontrolled phase Ib-II clinical trial in which a total of 20 patients ≥ 1 year of age with an allogeneic transplant of hematopoietic progenitors and post-transplant CMV infection will be included. The main objective is to evaluate the safety of the infusion of CMV activated T-lymphocytes and secondary objectives are to evaluate the efficacy through clinical evolution, viral load, ability to induce immunoreconstitution against the virus and evaluation of the persistence of specific T cells.

The treatment will be administered intravenously (central or peripheral route) in a single dose at a dose of 0.01-5 E4 specific virus T lymphocytes per Kg of receptor weight. After the infusion, patients will follow periodic controls (+7, +14, +21, +28, +45 and +60 days) in which a clinical evaluation will be performed and blood samples will be obtained in order to evaluate the persistence of specific T cells in the recipient:

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of an allogeneic hematopoietic progenitors cell transplant (irrespectively of the donor source, donor type conditioning and underlying disease) that is beyond the day +30 of the procedure
2. Patient with post-transplant infection due to CMV refractory or resistant to optimal pharmacological treatment. Specifically, the patient must be included in any of the following cases

   1. Patient with organic disease caused by CMV (confirmed by histology) resistant to antiviral first line treatment
   2. Patient with CMV reactivation and no organic disease, resistant or intolerant to 2 previous antiviral treatment lines (ganciclovir/valganciclovir and foscarnet) or not candidate to be treated due to not acceptable expected toxicity (severe renal insufficiency, neutropenia or severe thrombopenia) It is agreed that the patient is affected with a resistant CMV infection if the CMV copies doesn't decrease in > 1 log in total blood or otherwise the absolute number of copies > 1x10E4/mL in total blood after 2 weeks of antiviral treatment.
   3. Patients with reactivation of recurrent CMV despite correct anti-CMV treatment. It will be considered a recurrent CMV infection if the patient has > 2 reactivations in a period <6 months despite having received correct anti-CMV treatment
   4. Documented genetic mutations associated with ganciclovir or foscarnet resistance
3. ≥ 1 year of age
4. Estimated life expectancy > 30 days
5. Signature of the informed consent form

Exclusion Criteria:

1. Acute graft-versus-host disease (GVHD) ≥ grade II or chronic ≥ moderate
2. Corticosteroid ≥ 0.5mg/kg regardless the indication
3. Disease relapse at the time of infection or at any time after the Allogeneic transplant.
4. Severe renal disease (creatinine > 3gr/dL)
5. Severe hepatic disease (bilirubin >3mg/dL or aspartate aminotransferase (AST) >500 U/L) except if it is secondary to the viral infection.
6. Having received a donor lymphocytes infusion or any cell therapy product within 60 days prior to inclusion in the study (with the exception of transfusions), or having it planned within the next 60 days.
7. Alteration of the general condition, infection or clinical or hemodynamic instability that, in the opinion of the researcher, does not recommend the use of T cells
8. Known hypersensitivity to murine proteins or iron dextran.
9. Positive serology to human immunodeficiency virus (HIV), hepatitis B virus (HBV) (HBsAg, HBcAc), hepatitis C virus (HCV) and/or syphilis
10. Pregnant, lactating or women without adequate contraception
11. Participation in a clinical trial with investigational medicinal products the last 30 days

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Safety assessment: Adverse events | 60 days
  Adverse events

SECONDARY OUTCOMES:
Polymerase chain reaction (PCR) | +7, +14, +21, +28, +45, +60 days
  Quantitative viral load
IFN-γ+ spot forming cells | +7, +14, +28, +60 days
  Immune reconstitution by Elispot
Lymphocyte subpopulations | +7, +14, +28, +60 days
  Immune reconstitution by flow cytometry
T-cell persistence by chimerism | +14, +28 days
  Detection of donor cellularity (administered product) in the receptor serum
Time elapsed in identifying the donor | Day 0
  Time elapsed between the patient's inclusion in the trial and confirmation of the donor

CONTACTS AND LOCATIONS:
Overall Officials: Pere Barba, MD, PhD, Principal Investigator — VHIO (Vall d'Hebron Institute of Oncology)
Locations (7):
- Spain (7):
  - ICO Badalona, Badalona, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - ICO l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Blood and Tissue Bank of Catalonia — http://www.bancsang.net
- See also: Vall d'Hebron Institute of Oncology — http://www.vhio.net